CLINICAL TRIAL: NCT06865937
Title: Context-Aware Mobile Intervention for Social Recovery in Serious Mental Illness (R33)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Granholm, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33MH126094 (NIH); 4R33MH126094-03 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Schizophenia Disorder; Schizoaffective Disorder
Keywords: schizophrenia; serious mental illness; social engagement; randomized clinical trial
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile Social Interaction Therapy by Exposure (mSITE) (Experimental): mSITE is a blended intervention that integrates a brief in-person psychotherapy with context-triggered mobile smartphone intervention and remote telephone coaching.
  Interventions: Behavioral: Mobile Intervention for Social Recovery in Serious Mental Illness (mSITE)
- Supportive Contact (SC) (Active Comparator): The SC arm is a contact condition that will provide the same amount of individual in-person and coaching, and mobile device contact as the mSITE condition.
  Interventions: Behavioral: Supportive Contact (SC)

INTERVENTIONS:
Behavioral: Mobile Intervention for Social Recovery in Serious Mental Illness (mSITE) — mSITE is a blended intervention that integrates a brief in-person psychotherapy with context-triggered mobile smartphone intervention and remote telephone coaching. Participants will attend weekly, in-person sessions for 8 weeks and then 15-minute, remote coaching sessions for 10 weeks. The intervention begins with setting a meaningful recovery goal and then the generic cognitive model is introduced and a simple thought challenging skill is trained to specifically address social avoidance behaviors and facilitate work toward recovery goals. Defeatist attitudes, social threat and avoidance behaviors that interfere with working on the goal are then modified using cognitive-behavioral therapy skills and practiced using role-plays.
  Arms: mobile Social Interaction Therapy by Exposure (mSITE)
Behavioral: Supportive Contact (SC) — The SC arm will match the mSITE arm on the same amount of individual in-person and coaching, and mobile device contact. Coaching sessions will be semi-structured and consist of setting recovery goals, check-in about symptoms and potential crisis management, flexible discussion involving psychoeducation, instructions for accessing community crisis lines and community resources, and symptom management behaviors that grow out of discussions, with only minimal therapist guidance.
  Arms: Supportive Contact (SC)

SUMMARY:
This randomized clinical trial will test a new technology-supported blended intervention, mobile Social Interaction Therapy by Exposure (mSITE), that targets social engagement in consumers with serious mental illness.

DETAILED DESCRIPTION:
This study evaluates a new technology-supported blended intervention, mobile Social Interaction Therapy by Exposure (mSITE), that targets social behavior, and it also validates several new techniques for measuring social behavior. mSITE blends brief in-person psychotherapy with a context-triggered mobile smartphone intervention and remote telephone coaching. The investigators will conduct a randomized clinical trial of mSITE, evaluating whether the intervention leads to clinically significant changes in the frequency of social interactions in comparison to a therapist and device matched condition. The investigators will changes in outcome measures at baseline and Weeks 8, 18, and 30. If found to be effective, a scalable intervention that reduces social isolation in serious mental illness would have significant personal, societal, and economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent to participate and capacity to consent; Age 18 to 65;
* Diagnosis of schizophrenia, schizoaffective, bipolar I disorder or major depression with history of psychosis based on a diagnostic interview and available medical record review;
* Minimum level of social avoidance defined by a score of ≥ 2 on the Scale for the Assessment of Negative Symptoms (SANS) asociality item;
* Be willing and able to speak English at ≥ 6th grade reading level (to read intervention workbook).

Exclusion Criteria:

* Prior cognitive-behavioral therapy in the past 2 years;
* Greater than moderate disorganization on the PANSS (P2- Disorganization item >5);
* Alcohol or substance dependence in past 3 months based on the diagnostic interview;
* Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness);
* Unable to adequately see or manually manipulate a phone;
* Resident of an integrated housing facility that also provides treatment services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment | Assess change from baseline in number of social interactions at Weeks 0, 8, 18, and 30.
  Ecological Momentary Assessment (EMA) is a method of remote data collection that involves repeatedly sampling a participant's current behaviors, thoughts, mood, and experiences in real time, in their natural environments. The primary outcome in this study will be the number of social interactions.
Clinical Assessment Interview for Negative Symptoms | Assess change from baseline in number of social interactions at Weeks 0, 8, 18, and 30.
  Measure changes in motivational negative symptoms on the Clinical Assessment Interview for Negative Symptoms (CAINS). The CAINS is a 13-item interview-based assessment of negative symptoms, and each item is rated from 0 (no impairment) to 4 (severe deficit) measuring the two negative symptom factors recommended in consensus reports: Expression and Motivation and Pleasure (MAP) across social, vocational and recreational domains. Total scores for each factor are computed. The range for the MAP is 0 - 36, and the range for the Expression factor is 0 - 16. Higher scores indicate more severe negative symptoms for both factors.
Birchwood Social Functioning Scale | Assess change from baseline in number of social interactions at Weeks 0, 8, 18, and 30.
  Measure changes in functioning on the Birchwood Social Functioning Scale (SFS). The SFS is a self-report assessment of functioning with 7 subscales, and each item is rated from 0 to 3 with the exception of the Occupation/Employment subscale if a participant is in regular employment (scores range from 7-10 based upon type of work). The subscales and score ranges are: Social Engagement Withdrawal (0-15), Interpersonal Communication/Relationships (0-30), Prosocial Activities (0-66), Recreation (0-48), Independence-Performance (0-39), Independence-Competence (0-39), and Occupation/Employment (0-10). Higher scores indicate better functioning for all subscales.
Positive And Negative Syndrome Scale | Assess change from baseline in number of social interactions at Weeks 0, 8, 18, and 30.
  The Positive And Negative Syndrome Scale (PANSS) is a 30-item interview that provides balanced representation of positive and negative symptoms and gauges their relationship to one another and to global psychopathology. Items are rated 1 (Absent) to 7 (Extreme) and summed across items for a total range of scores of 30-210. Higher scores indicate the presence of more severe symptoms.
Passive sensing mobile application | Assess change from baseline in number of social interactions at Weeks 0, 8, 18, and 30.
  The passive sensing mobile application will measure the number of conversations. The conversations or specific content will not be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Granholm, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California - San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Per terms of the award, participant-level data will be uploaded to the NIMH Data Archive (NDA).
Time Frame: Data will be uploaded according to NDA standard data submission periods. These periods are currently twice each year.
Access Criteria: Data access is outlined in the current NDA Policy.
URL: https://nda.nih.gov/